CLINICAL TRIAL: NCT02372747
Title: Comparison of Delta-Shaped and Billroth II for Intracorporeal Anastomosis After Totally Laparoscopic Distal Gastrectomy for Gastric Cancer
Brief Title: Comparison of Delta-Shaped and Billroth II After TLDG
Acronym: TLDG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Deputy Director of General Surgery, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013-179
Record Dates: First submitted 2015-01-22; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2006-02

CONDITIONS: Gastric Cancer
Keywords: Totally laparoscopic gastrectomy; laparoscopic distal gastrectomy; Intracorporeal anastomosis; Delta-Shaped Anastomosis; Billroth II Anastomosis; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delta-shaped anastomosis group (Experimental): The patients in DS group underwent Delta-shaped anastomosis after TLDG.
  Interventions: Procedure: Delta-shaped anastomosis
- Billroth II anastomosis group (Experimental): The patients in B-II group underwent Billroth-II anastomosis after TLDG.
  Interventions: Procedure: Billroth II anastomosis

INTERVENTIONS:
Procedure: Delta-shaped anastomosis — The patients in DS group underwent Delta-shaped anastomosis after TLDG.
  Arms: Delta-shaped anastomosis group
Procedure: Billroth II anastomosis — The patients in B-II group underwent Billroth-II anastomosis after TLDG.
  Arms: Billroth II anastomosis group

SUMMARY:
To compare the safety and feasibility of Delta-shaped anastomosis and Billroth II anastomosis after totally laparoscopic distal gastrectomy for gastric cancer(TLDG).

DETAILED DESCRIPTION:
Methods: 78 consecutive patients who underwent TLDG in First Hospital of Jilin University between October 2012 and December 2014 were enrolled in this study . All patients were divided randomly into two groups:Delta-shaped anastomosis group (DS group) and Billroth II anastomosis group (B-II group), and the patients in DS group underwent Delta-shaped anastomosis after TLDG, and the patients in B-II group underwent Billroth-II anastomosis after TLDG.Outcome measures,resected margin,operative time,anastomosis time,number of stapler cartridges used,length of the incision,the time of first flatus and liquid diet,hospital stay and postoperative morbidity are compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* carcinoma located in the lower 1/3 of gastric body or antrum of stomach
* diagnosed by endoscopy ,endoscopic ultrasonography and abdominal CT scan
* diameter of the tumor <3cm
* no pyloric obstruction

Exclusion Criteria:

* diameter of the tumor ≥3cm
* associated with obstruction, bleeding, emergency surgery or surgical intervention
* tumor with extensive metastasis
* patient had previously undergone gastrostomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Stage distribution | up to 7 days after the operation
Resected margin | up to 7 days after the operation
Operative time | up to 7 days after the operation
Anastomosis time | up to 7 days after the operation
The number of stapler cartridges used | up to 7 days after the operation
Median estimated blood loss | up to 7 days after the operation
Red blood cell transfusion | up to 7 days after the operation
Length of the incision | up to 7 days after the operation

SECONDARY OUTCOMES:
Postoperative complication | up to 30 days after the operation
  Major complications includes anastomosis leakage and intrabdominal bleeding . Minor complications includes bile regurgitation,anastomotic stenosis and delayed gastric emptying.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Wang, Doctor, Study Director — The First Hospital of Jilin University